CLINICAL TRIAL: NCT00367705
Title: Double-blind Placebo Controlled Trial of VSL#3 in Children With Crohn's Disease
Brief Title: VSL#3 Treatment in Children With Crohn's Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Prof. David Branski, Hadassah Medical Organization
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: VSL-HMO-CTIL
Record Dates: First submitted 2006-08-22; First posted 2006-08-23 (Estimated); Last update posted 2009-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- T (Active Comparator): VSL-#3
  Interventions: Dietary Supplement: VSL#3®
- P (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: VSL#3® — 1-2 sachets/day per os, 6 months
  Arms: T
Dietary Supplement: Placebo — 1-2 sachets/day per os, 6 months
  Other Names: placebo powder
  Arms: P

SUMMARY:
Crohn's disease (CD) in childhood is a chronic relapsing and remitting condition that has a significant impact on growth and development. The disease is characterized by an increased and unregulated immune response. The main therapy over the last 30 years has been corticosteroids leading to remission in 50-80% of patients within 2-4 weeks. However, the use of steroids in children is limited by side-effects including acne, moon-face, hirsutism, hypertension, metabolic disturbances and above all reduced growth. Hence, pediatricians are very interested to find alternative therapies. Therapeutic manipulation of gut flora with probiotics promises to be a useful strategy for several disorders including inflammation of the gut. The efficacy of the highly concentrated probiotic VSL#3 has been documented in maintenance and prophylaxis treatment of pouchitis in double blind, placebo controlled studies in adults. The aim of this study is to compare probiotic therapy with VSL#3 versus placebo in maintenance therapy of children with mild to moderate CD, treated with either 5-ASA, corticosteroids (local or budesonide), imuran/6 mercaptopurine (MP), as long as no change in medication dosage has been made in the previous 12 weeks (for imuran/6MP) or 4 weeks (for corticosteroids).

DETAILED DESCRIPTION:
The aim of this study is to compare probiotic therapy with VSL#3 versus placebo in maintenance therapy of children with mild to moderate CD, treated with either 5-ASA, corticosteroids (local or budesonide), imuran/6MP, as long as no change in medication dosage has been made in the previous 12 weeks (for imuran/6MP) or 4 weeks (for corticosteroids). The primary goal will be to compare their ability to maintain remission and to decrease disease activity in each of the two study groups. Data will be collected during this 16 week period regarding the safety and tolerability of VSL#3, as well as data of changes in stool composition of microflora upon treatment.

The follow up will be continued for up to 6 months with a monthly telephone questionnaire and a clinical visit at 6 months.

Study Design:

The study will be a multinational, double-blind, randomized controlled study (Munich, Paris, Rotterdam, Porto, Brussels, London, Warsaw, Chicago, Toronto, Boston, New York, Baltimore, Cleveland, Karachi and Jerusalem).

The study will include 300 children and will last for at least 16 weeks. These children will receive either 1-2 packet according to their weight; each sachet containing 900 billion bacteria/day of VSL#3 or an identical placebo, for 16 weeks.

All patients participating in this study will continue regular medications throughout the study period.

According to the Pediatric Crohn's Disease Activity Index (PCDAI) patients will be assessed clinically at regular intervals and will have stool cultured (including lactobacillus, bifidobacteria and Strep salivarius) as well as a stool calprotectin before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 6 - 18 years
2. Previous diagnosis of Crohn's disease or newly diagnosed with symptoms for at least three months before recruitment to the study.The diagnosis of CD is established by:

   1. history and symptoms of the disease
   2. endoscopy/histology or radiology with negative stool culture.
3. Written informed consent by parent
4. PCDAI > 12.5 and < 30
5. Treatment with 5-ASA, budesonide and imuran/6MP daily provided that the dose has remained stable for the 4 weeks (corticosteroids) or 12 weeks (for imuran/6MP) prior to inclusion. Children treated with other medications (such as anti-TNF or antibiotics including ciprofloxacilin or metronidazole) cannot enter this study.

Exclusion Criteria:

1. Short bowel syndrome/ileostomy/abscess/fistula/small bowel obstruction/stenosis/stricture
2. Imminent surgery
3. Treatment with anti-TNF, systemic corticosteroids, ciprofloxacillin, metronidazole within 12 weeks of the start of the trial.
4. Participation in another clinical trial within the last 30 days.
5. Patients should not take antibiotics during the study.
6. Patients should not take opioids, cholestyramine, ursodeoxycholic acid during the study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-09 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
remission | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: David Branski, MD, Study Director — Hadassah Medical Organization; Michael Wilschanski, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization,, Jerusalem, Israel

REFERENCES:
- [Background] Gionchetti P, Rizzello F, Lammers KM, Morselli C, Sollazzi L, Davies S, Tambasco R, Calabrese C, Campieri M. Antibiotics and probiotics in treatment of inflammatory bowel disease. World J Gastroenterol. 2006 Jun 7;12(21):3306-13. doi: 10.3748/wjg.v12.i21.3306. PMID 16733845